CLINICAL TRIAL: NCT03093012
Title: Individual Blood Pressure Optimization Based on Cerebral Blood Flow Autoregulation After Implantation of Continuous-flow Left Ventricular Assist Device
Brief Title: Individual Blood Pressure Optimization Based on Cerebral Autoregulation After Implantation of Continuous-flow LVAD
Acronym: NIRS
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: International Society for Heart and Lung Transplantation (Other)
Responsible Party: Principal Investigator, Kenneth Liao, Principal Investigator, Baylor College of Medicine
Other Study IDs: H-34866
Record Dates: First submitted 2017-02-22; First posted 2017-03-28 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Heart-Assist Devices; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will collect retrospective and prospective clinical data regarding the Principal Investigator's patient population to allow for data analysis seeking basic trends and to prepare academic reports, including journal manuscripts and presentations for scientific organizations.

DETAILED DESCRIPTION:
Preoperative data will be collected as the baseline information through chart review and patient interview before the surgery as follows: patient demographics, co-morbidities, medication, preoperative laboratory results, and preoperative vital signs.

Intraoperative data will be collected by chart review or monitor review as follows: type of implant device, concomitant procedures, length of surgery, duration of cardiopulmonary bypass and aortic cross clamp, blood products administered hemodynamic variables, and NIRS signals.

Postoperative data will be collected by chart review or monitor review as follows: medications, blood products administered, postoperative laboratory results, adverse events and operative mortality*, length of mechanical ventilation, length of inotrope administered, hemodynamic variables, length of intensive care unit and hospital stay, mortality, and NIRS signals.

Participants will receive routine standard institutional perioperative care that included invasive radial artery blood pressure monitoring. Participants will be connected to the NIRS monitor using sensor probes placed on the right and left sides of the forehead per routine clinical application. NIRS signal monitoring will be initiated before induction of general anesthesia in the operation room for collecting baseline data, and continued during LVAD implantation procedure. After implantation of LVAD, continuous NIRS monitoring will be carried out in the ICU until termination of the invasive arterial blood pressure monitoring.

For all participants enrolled in this study, all medical treatment which is provided will not deviate from the standard of clinical care, including surgery and other procedures as well as blood sample collection. The data will be reviewed routinely to seek trends. When needed to examine specific clinical issues, such as risk factors for a given complication, additional clinical data will be retrieved from the medical records. All data sets analyzed and used for presentations or publication will be anonymized to protect patient confidentiality. This study will be conducted indefinitely.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients greater than or equal to 18 years old undergoing continuous-flow left ventricular assist device implantation for the clinical indications of bridge to transplant or destination therapy.

Exclusion Criteria:

* Patients < 18 years of age will be ineligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects implanted with continuous-flow left ventricular assist device
Sampling Method: Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-03-07 (Actual); Study Completion 2018-03-07 (Actual)

PRIMARY OUTCOMES:
Individual optimal blood pressure change between before and after continuous-flow LVAD implantation determined by cerebral autoregulation monitoring with NIRS | From initiation of cerebral autoregulation monitoring in operation room until termination of the invasive arterial blood pressure monitoring in ICU (up to 48 hours)
  Using cerebral autoregulation monitoring method, the optimal blood pressure for maintaining cerebral blood flow (CBF) can be determined individually. The individual optimal blood pressure to maintain CBF autoregulation will be determined and assessing change between before and after implantation of continuous-flow LVAD.

SECONDARY OUTCOMES:
Extent of impairment of cerebral autoregulation in perioperative periods | From initiation of cerebral autoregulation monitoring in operation room until termination of the invasive arterial blood pressure monitoring in ICU (up to 48 hours)
  Using cerebral autoregulation monitoring method, the extent of impairment of cerebral autoregulation can be determined (AUCMAP: area under the curve of excursion of mean arterial pressure), which is calculated with magnitude (mmHg) and duration (hour) of mean arterial pressure (MAP) excursions below the individual optimal blood pressure to maintain cerebral autoregulation.
Postoperative adverse events and operative mortality after continuous-flow LVAD implantation. | From implantation of continuous-flow LVAD until discharge of hospital (up to 4 weeks)
  Postoperative adverse events including followings: 1) stroke; persistent neurological deficit >24 hours, 2) renal failure; new requirement for dialysis postoperatively or increase in creatinine to >2 mg/dL and 2 times greater than baseline, acute kidney injury; RIFLE criteria, 3) respiratory failure; mechanical lung ventilation >72 hours or requirement for tracheotomy, 4) right ventricular failure; requirement for right ventricular assist device, 5) operative mortality; all deaths that occur during the hospitalization in which the operation is performed, even if after 30 days, and deaths that occur after discharge from the hospital but within 30 days of the procedure, unless the cause of death was clearly unrelated to the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Masahiro Ono, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will collect retrospective and prospective clinical data regarding the Principal Investigator's patient population to allow for data analysis seeking basic trends and to prepare academic reports, including journal manuscripts and presentations for scientific organizations.

REFERENCES:
- [Background] Brady K, Joshi B, Zweifel C, Smielewski P, Czosnyka M, Easley RB, Hogue CW Jr. Real-time continuous monitoring of cerebral blood flow autoregulation using near-infrared spectroscopy in patients undergoing cardiopulmonary bypass. Stroke. 2010 Sep;41(9):1951-6. doi: 10.1161/STROKEAHA.109.575159. Epub 2010 Jul 22. PMID 20651274
- [Background] Brady KM, Lee JK, Kibler KK, Smielewski P, Czosnyka M, Easley RB, Koehler RC, Shaffner DH. Continuous time-domain analysis of cerebrovascular autoregulation using near-infrared spectroscopy. Stroke. 2007 Oct;38(10):2818-25. doi: 10.1161/STROKEAHA.107.485706. Epub 2007 Aug 30. PMID 17761921
- [Background] Ono M, Joshi B, Brady K, Easley RB, Kibler K, Conte J, Shah A, Russell SD, Hogue CW. Cerebral blood flow autoregulation is preserved after continuous-flow left ventricular assist device implantation. J Cardiothorac Vasc Anesth. 2012 Dec;26(6):1022-8. doi: 10.1053/j.jvca.2012.07.014. PMID 23122299
- [Background] Ono M, Brady K, Easley RB, Brown C, Kraut M, Gottesman RF, Hogue CW Jr. Duration and magnitude of blood pressure below cerebral autoregulation threshold during cardiopulmonary bypass is associated with major morbidity and operative mortality. J Thorac Cardiovasc Surg. 2014 Jan;147(1):483-9. doi: 10.1016/j.jtcvs.2013.07.069. Epub 2013 Sep 26. PMID 24075467
- [Background] Ono M, Arnaoutakis GJ, Fine DM, Brady K, Easley RB, Zheng Y, Brown C, Katz NM, Grams ME, Hogue CW. Blood pressure excursions below the cerebral autoregulation threshold during cardiac surgery are associated with acute kidney injury. Crit Care Med. 2013 Feb;41(2):464-71. doi: 10.1097/CCM.0b013e31826ab3a1. PMID 23263580
- [Background] Aries MJ, Czosnyka M, Budohoski KP, Steiner LA, Lavinio A, Kolias AG, Hutchinson PJ, Brady KM, Menon DK, Pickard JD, Smielewski P. Continuous determination of optimal cerebral perfusion pressure in traumatic brain injury. Crit Care Med. 2012 Aug;40(8):2456-63. doi: 10.1097/CCM.0b013e3182514eb6. PMID 22622398
- [Background] Lee JK, Kibler KK, Benni PB, Easley RB, Czosnyka M, Smielewski P, Koehler RC, Shaffner DH, Brady KM. Cerebrovascular reactivity measured by near-infrared spectroscopy. Stroke. 2009 May;40(5):1820-6. doi: 10.1161/STROKEAHA.108.536094. Epub 2009 Mar 12. PMID 19286593